CLINICAL TRIAL: NCT00262275
Title: Optimum Platelet Inhibition After Coronary Artery Bypass Surgery: A Randomised Trial Comparing Platelet Aggregation Using Low, Medium Dose Aspirin and Clopidogrel
Brief Title: Optimum Platelet Inhibition After Coronary Bypass Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Papworth Hospital NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LREC 01/624
Record Dates: First submitted 2005-12-05; First posted 2005-12-06 (Estimated); Last update posted 2016-01-22 (Estimated); Status verified 2016-01

CONDITIONS: Ischemic Heart Disease
MeSH Terms: conditions — Myocardial Ischemia | interventions — Aspirin; Clopidogrel

INTERVENTIONS:
Drug: Aspirin, Clopidogrel

SUMMARY:
To investigate the effect of different dosages of aspirin on platelet aggregation and to determine the possible mechanisms of aspirin resistance, we intend to compare the effects of low, medium dose aspirin with clopidogrel (an alternative antiplatelet agent) in patients after coronary artery bypass surgery.

ELIGIBILITY:
Inclusion Criteria:

We intend to invite patients aged 18 to 80 proceeding to primary elective coronary artery bypass surgery, able to give informed consent.

Exclusion Criteria:

Preoperative exclusion criteria:

* patients who are have not stopped aspirin 7 days prior to surgery
* patients on concomitant NSAIDS
* patients with a previous history platelet disorders, splenectomy or haematological disorders
* patients with aspirin induced asthma
* patients with any contraindications to aspirin (GI bleed)
* patients who are on any medication that may result in a serious drug interaction with aspirin (warfarin)
* Women of childbearing potential
* Patients of less than 18 years
* If informed consent cannot be obtained
* If for any reason the consultant surgeon or anaesthetist deems it to be appropriate

Operative exclusion criteria:

• Concomitant procedures

Postoperative exclusion criteria:

* patients who receive platelet transfusion
* patients who receive NSAIDS
* requirement for intra aortic balloon pump support
* failure of extubation within 24 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-07; Primary Completion 2004-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Lim, MB ChB, MSc, MRCS, Principal Investigator — Papworth Hospital NHS Foundation Trust
Locations (1):
- Papworth Hospital, Cambridge, United Kingdom

REFERENCES:
- [Result] Lim E, Cornelissen J, Routledge T, Kirtland S, Charman SC, Bellm S, Munday H, Khan O, Masood I, Large S. Clopidogrel did not inhibit platelet function early after coronary bypass surgery: A prospective randomized trial. J Thorac Cardiovasc Surg. 2004 Sep;128(3):432-5. doi: 10.1016/j.jtcvs.2004.03.007. PMID 15354104
- [Result] Lim E, Cornelissen J, Routledge T, Ali A, Kirtland S, Sharples L, Sheridan K, Bellm S, Munday H, Large S. Biological efficacy of low versus medium dose aspirin after coronary surgery: results from a randomized trial [NCT00262275]. BMC Med. 2006 May 22;4:12. doi: 10.1186/1741-7015-4-12. PMID 16716214
- [Derived] Lim E, Carballo S, Cornelissen J, Ali ZA, Grignani R, Bellm S, Large S. Dose-related efficacy of aspirin after coronary surgery in patients With Pl(A2) polymorphism (NCT00262275). Ann Thorac Surg. 2007 Jan;83(1):134-8. doi: 10.1016/j.athoracsur.2006.08.002. PMID 17184645